CLINICAL TRIAL: NCT06017219
Title: Bioavailability of Spermidine in Healthy Males
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chrysea Labs Lda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AFCRO 167
Record Dates: First submitted 2023-08-14; First posted 2023-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Spermidine

STUDY DESIGN:
Intervention Model Description: single blind cross over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- within subject control 20mg (Experimental): spermidine
  Interventions: Dietary Supplement: spermidine
- within subject control 40mg (Experimental): spermidine
  Interventions: Dietary Supplement: spermidine

INTERVENTIONS:
Dietary Supplement: spermidine — spermidine

SUMMARY:
To evaluate in healthy males the safety of two doses of spermidine as assessed by occurrence of any Adverse Events/Serious adverse events.

DETAILED DESCRIPTION:
Until now, lack of availability of a reproducible high quality, uncontaminated, spermidine for human consumption as a food or supplement has been a significant barrier to its study and use.

Chrysea is producing spermidine by a patented biological process to consistently produce very high purity spermidine to pharmaceutical and food grade standards.

Using a rat ex vivo jejunal absorption model and 14Carbon labelled spermidine, the recovery rate of radioactivity at the portal vein was approximately 61-76% during the initial 10 minutes after the administration of 14C-spermidine.

Data on spermidine absorption in humans is very limited. The purpose of this single blind randomised pharmacokinetic study is to demonstrate absorption of 20mg and 40 mg doses of spermidine in fasted normal volunteers, and to describe the absorption kinetics (Tmax, Cmax, T1/2, AUC).

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent.
* Male.
* Age between 18-70 years inclusive.
* BMI between ≥18.5 and ≤28 kg/m2.
* In general good health, as determined by the investigator.
* Agree to abstain from consuming alcohol, grapefruit, or grapefruit juice for 72 hours prior to visit 2 and visit 3.
* Adequate vein access for cannulation and multiple blood draws.
* Able to communicate well with the Investigator, to understand and comply with the requirements of the study and be judged suitable for the study in the opinion of the Investigator.
* Willing to consume the study product.

Exclusion Criteria:

* History of anaphylaxis,
* Documented hypersensitivity reaction or a clinically important reaction to any dietary/food supplement or drug,
* Intolerance or sensitivity to study product ingredients

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Cmax. To evaluate the pharmacokinetics of two different doses (20 mg and 40mg) of spermidine in healthy males | Pre dosing to dosing plus six hours
  Maximum concentration of circulating spermidine (Cmax)
Tmax. To evaluate the pharmacokinetics of two different doses (20 mg and 40mg) of spermidine in healthy males | Pre dosing to dosing plus six hours
  Time to peak of circulating spermidine (Tmax)
T 1/2. To evaluate the pharmacokinetics of two different doses (20 mg and 40mg) of spermidine in healthy males. | Pre dosing to dosing plus six hours
  Half-life of circulating spermidine (t1/2)
AUC. To evaluate the pharmacokinetics of two different doses (20 mg and 40mg) of spermidine in healthy males | Pre dosing to dosing plus six hours
  Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Patrick Keohane, Study Director — Chrysea Labs
Locations (1):
- Atlantia Clinical Trials, 1st Floor, Block C, Heron House, Blackpool Retail Park, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uda K, Tsujikawa T, Fujiyama Y, Bamba T. Rapid absorption of luminal polyamines in a rat small intestine ex vivo model. J Gastroenterol Hepatol. 2003 May;18(5):554-9. doi: 10.1046/j.1440-1746.2003.03020.x. PMID 12702048